CLINICAL TRIAL: NCT05118100
Title: Effectiveness of Adhesive Containing MDPB: a Practice-based Clinical Trial
Brief Title: Effectiveness of Adhesive Containing MDPB
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021THKHOLL01
Record Dates: First submitted 2021-10-27; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Secondary Caries
MeSH Terms: interventions — Clearfil Protect Bond; Clearfil SE Bond

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Protect Bond: Restoration placed using Clearfil Protect Bond adhesive (Kuraray Noritake, Osaka, Japan) , which contains the antibacterial monomer MDPB (12-Methacryloyloxydodecylpyridiniumbromide)
  Interventions: Drug: Clearfil Protect Bond
- SE Bond: Restoration placed using Clearfil SEBond adhesive (Kuraray Noritake, Osaka, Japan)
  Interventions: Drug: Clearfil SE Bond

INTERVENTIONS:
Drug: Clearfil Protect Bond — An adhesive is used routinely when placing resin composite restorations. This group receives a commercially available adhesive containing an antibacterial monomer (MDPB)
  Other Names: 12-Methacryloyloxydodecylpyridiniumbromide
  Groups: Protect Bond
Drug: Clearfil SE Bond — An adhesive is used routinely when placing resin composite restorations. This group receives a commercially available adhesive.
  Groups: SE Bond

SUMMARY:
9 general practices in the Netherlands were provided with two composite resin adhesives, each for a period of 9 months. One contained MDPB (Adhesive P), and the other one was used as a control (Adhesive S). Patient's age, SES, and caries risk, as well as tooth type/number, reason for restoration placement, used restorative material and bonding agent, and affected surfaces were recorded. All interventions carried out on these teeth in the next 6 years were extracted from the electronic patient records, along with their date, type, reason, and surfaces. Two dependent variables were defined: general failure, and failure due to secondary caries. All data handling and statistical analyses were carried out in R 4.0.5.

ELIGIBILITY:
Inclusion Criteria:

* Needing at least one dental restoration

Exclusion Criteria:

* Opted out of data collection

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visited one of the participating general dental practices during the study period needing at least one dental restoration
Sampling Method: Non-Probability Sample
Enrollment: 5102 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Restoration survival | up to 5 years
  Time in years restoration has survived without needing dental re-intervention

SECONDARY OUTCOMES:
Failure through caries | up to 5 years
  Incidence of secondary caries leading to replacement of the restoration

IPD SHARING:
Plan to Share IPD: Yes
Anonimized data will be published in the DANS-easy archive. The study description are available to anyone, and the data are available upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available upon study publication.
Access Criteria: Any individual requesting access through the archive will obtain access
URL: https://easy.dans.knaw.nl/ui/home

REFERENCES:
- [Derived] Hollanders ACC, Kuper NK, Bronkhorst EM, Laske M, Huysmans MCDNJM. Effectiveness of adhesive containing MDPB: A practice-based clinical trial. Dent Mater. 2023 Aug;39(8):756. doi: 10.1016/j.dental.2023.06.011. Epub 2023 Jul 1. PMID 37394389